CLINICAL TRIAL: NCT01820637
Title: Stenting of the Superficial Femoral and/or Proximal Popliteal Artery Project With Boston Scientific's Innova Drug Eluting Stent
Brief Title: Stenting of the Superficial Femoral and/or Proximal Popliteal Artery Project
Acronym: MAJESTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2049
Record Dates: First submitted 2013-03-22; First posted 2013-03-29 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Atherosclerosis of Native Arteries of the Extremities
Keywords: atherosclerosis; SFA; PPA; lower extremities; stenting; paclitaxel
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test device arm (DES SFA) (Experimental): Patients in this arm will receive the study device: the Boston Scientific DES SFA Paclitaxel-Eluting Self-Expanding Stent System (DES SFA)
  Interventions: Device: The Boston Scientific DES SFA Paclitaxel-Eluting Self-Expanding Stent System (DES SFA)

INTERVENTIONS:
Device: The Boston Scientific DES SFA Paclitaxel-Eluting Self-Expanding Stent System (DES SFA) — Drug-eluting SFA self-expanding stent

SUMMARY:
To determine whether the Boston Scientific nitinol drug-eluting stent shows acceptable performance at 9 months when treating Superficial Femoral (SFA) and/or Proximal Popliteal Artery (PPA) lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 and older
* Subject (or Legal Guardian if applicable) has signed the consent form and is willing and able to provide consent before any study-specific tests or procedures are performed and agrees to attend all required follow-up visits
* Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4
* Stenotic, restenotic (from angioplasty only, previous treatment with drug coated balloon is not allowed) or occlusive lesion(s) located in the native superficial femoral artery or proximal popliteal artery:

  1. Degree of stenosis ≥70% by visual angiographic assessment
  2. Vessel diameter ≥ 4 and ≤ 6mm
  3. Total lesion length (or series of lesions) ≥30 mm and ≤110 mm

     * (Note: tandem lesions may be treated, provided that the tandem lesion segment can be covered with only one stent)
  4. Target lesion located at least three centimeters above the inferior edge of the femur
* Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08-23 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Müller-Hülsbeck, Prof., Principal Investigator — Ev. Luth. Diakonissenanstalt Flensburg
Locations (13):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown
  - Prince of Wales Hospital, Randwick
- Allgemeines Krankenhaus AKH, Vienna, Austria, Austria
- Belgium (3):
  - AZ Sint-Blasius, Dendermonde
  - Ziekenhuis Oost Limburg, Genk
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Germany (4):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen GmbH, Bad Krozingen
  - Ev. Luth. Diakonissenanstalt Flensburg, Flensburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universität Leipzig, Leipzig
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Braemar Hospital, Hamilton
  - Middlemore Hospital, Otahuhu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Derived] Muller-Hulsbeck S, Keirse K, Zeller T, Schroe H, Diaz-Cartelle J. Twelve-Month Results From the MAJESTIC Trial of the Eluvia Paclitaxel-Eluting Stent for Treatment of Obstructive Femoropopliteal Disease. J Endovasc Ther. 2016 Oct;23(5):701-7. doi: 10.1177/1526602816650206. Epub 2016 May 18. PMID 27193308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 57 subjects enrolled at 14 investigative centers in Europe, Australia and New Zealand. The first subject was enrolled on 23 August 2013. Enrollment was completed on 03 March 2014, when the last subject was enrolled.
Groups:
- Test Device Arm (DES SFA, ELUVIA™): All patients in this arm were treated with the study device.
  The Boston Scientific DES SFA Paclitaxel-Eluting Self-Expanding Stent System (DES SFA, ELUVIA™)
Period: Overall Study
Arm/Group | Test Device Arm (DES SFA, ELUVIA™)
Started | 57
Completed | 54
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test Device Arm (DES SFA, ELUVIA™)
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 54
  Asian | 1
  Other | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 10
  Austria | 3
  Belgium | 19
  Australia | 4
  Germany | 21
General Medical History [Count of Participants; unit: Participants]
  History of Smoking | 50
  Current Diabetes Mellitus | 20
  History of Hyperlipidemia requiring medication | 36
  History of Hypertension requiring medication | 42
  History of Chronic Obstructive Pulmonary Disease | 6
  History of Coronary Artery Disease (CAD) | 22
  History of Myocardial Infarction (MI) | 9
  History of Congestive Heart Failure (CHF) | 3
  History of Percutaneous Coronary Intervention(PCI) | 11
  History of Coronary Artery Bypass Graft (CABG) | 8
  Stable Angina | 6
  History of Transient Ischemic Attacks (TIA) | 3
  History of Cerebrovascular Accident (CVA) | 5
  History of Renal Insufficiency | 5
  History of Renal Percutaneous Intervention | 1
  History of Peripheral Vascular Surgery | 3
  History of Peripheral Endovascular Intervention | 14
  History of Claudication | 51

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Primary patency of target lesion at 9-months assessed by duplex ultrasound (DUS) as adjudicated by an independent core laboratory. Primary Patency: percentage (%) of lesions (target stented segments) that reach endpoint without a hemodynamically significant stenosis on DUS and without target lesion revascularization (TLR) or, bypass of the target lesion.
Time Frame: 9-months
Population: 54 subjects were included in this analysis - one 9 month visit was completed too early, outside the protocol defined visit window, one subject withdrew consent at the 1 month follow-up visit and one subject did not complete the 9 month follow up visit due to site relocation.
Measure: Number (90% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Test Device Arm (DES SFA, ELUVIA™)
Number analyzed (Participants) | 54
Number analyzed (Lesions) | 54
percentage of lesions | 94.4 [86.3 to 98.5]

2. Other Pre Specified Outcome: Percentage of Participants With Composite of Major Adverse Events
Description: The composite rate of Major Adverse Events (MAEs) is defined as all causes of death through 1 month, target limb major amputation through 9 months and/or target lesion revascularization through 9 months.
Time Frame: 9 months
Population: 55 subjects were included in this analysis - one subject withdrew consent at the 1 month follow-up visit and one subject did not complete the 9 month follow up visit due to site relocation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Test Device Arm (DES SFA, ELUVIA™)
Number analyzed (Participants) | 55
percentage of participants
  9-Month MAE (Composite Endpoint) | 3.6 [0.4 to 12.5]
  All Causes of Death at 1 month | 0.0 [0.0 to 6.5]
  Target Limb Major Amputation | 0.0 [0.0 to 6.5]
  Target Lesion Revascularization (TLR) | 3.6 [0.4 to 12.5]

ADVERSE EVENTS:
Time Frame: 3 years +/- 30 days visit window from the date of the index procedure.
Arm/Group | Test Device Arm (DES SFA, ELUVIA™)
All-Cause Mortality (participants affected / at risk) | 2/57
Serious Adverse Events (participants affected / at risk) | 34/57
Other Adverse Events (participants affected / at risk) | 36/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Device Arm (DES SFA, ELUVIA™) (N=57)
Femoral artery stenosis (Vascular disorders) | 14 (21)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (6)
Arterial thrombosis limb (Vascular disorders) | 3 (5)
Arterial stenosis limb (Vascular disorders) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 1 (3)
Femoral artery occlusion (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arterial spasm (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Cardiac death (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Device Arm (DES SFA, ELUVIA™) (N=57)
Femoral arterial stenosis (Vascular disorders) | 9 (13)
Femoral artery occlusion (Vascular disorders) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 2 (2)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3)
Catheter site haematoma (General disorders) | 2 (3)
Catheter site haemorrhage (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 3 (3)
Feeling cold (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 2 (2)
Abnormal sensation in eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Hyphaema (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the Results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor from the proposed publication or presentation.